CLINICAL TRIAL: NCT02094313
Title: Effects of Decrease in Cholesterol Levels Induced by a Statin on Sperm Quality
Brief Title: Effects of Atorvastatin on Human Semen and Gonadal Hormones
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Service de Biologie de la Reproduction : AMP-CECOS (Unknown); EA 975, Laboratoire de BDR (Unknown); Service d'Endocrinologie, Diabète et Maladies Métaboliques (Unknown); Laboratoire d'Hormonologie - Biochimie (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0185; 2006-004376-12
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers; Normocholesterolaemic Men; Normozoospermic Men
Keywords: Atorvastatin; Human Spermatozoa; Seminal fluid; Accessory Glands; Cholesterol; Gonadotropins,; Testosterone
MeSH Terms: interventions — Atorvastatin; Anticholesteremic Agents

ARMS (1):
- atovastatin (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — The aim of this pilot study is to evaluate the efficacy and the safety of a decrease of cholesterol blood levels, induced by taking atorvastatin, on sperm quality of normocholesterolaemic and healthy men without confounding factors.
  Other Names: cholesterol lowering drug

SUMMARY:
Recently, concerns about the effect of atorvastatin intake on men fertility have been raised. However, this statin has never been investigated regarding its influence on male fertility, notably sperm quality.

The aim of this pilot study is to evaluate the efficacy and the safety of a decrease of cholesterol blood levels, induced by taking atorvastatin, on sperm quality of normocholesterolaemic and healthy men without confounding factors.

DETAILED DESCRIPTION:
The main objective is to estimate the safety of atorvastatin on fertility of normocholesterolaemic and healthy men (having normal blood lipid profile and normal sperm parameters) by analyzing its effects on sperm parameters: ejaculate volume, sperm count, total and progressive motility, percentage of typical forms.

The secondary objectives are to assess the changes in:

* hormonal profile: gonadotropins and testosterone plasma levels
* lipid composition of sperm and seminal fluid;
* spermatozoa capacitation markers
* accessory glands markers.

The efficacy is estimated by measuring the lipid lowering action of atorvastatin. It is expected a decrease by 20 and 40% of total cholesterol blood and LDL-cholesterol levels, respectively (total cholesterol <1.5 g / l and LDL-cholesterol <1g / l).

Considering this protocol as a pilot study to evaluate safety and efficacy, sample size estimation was fixed considering a Fleming design at one stage. These designs with one group and multi-stages (between 1 and 5) can be seen as filtering steps leading to the decision type go/no go. With a type I error a and statistical power (1-β) equals respectively 5% and 90%, n=17 subjects were necessary to reject the hypotheses of minimal (p=0.85) and maximal (p=0.95) acceptable non-toxicity. If 1 subject or more presented a toxicity, the treatment was considered no safe. To measure the evolution of total cholesterol and LDL-cholesterol levels concerning the efficacy, n=17 subjects were necessary to show a minimal paired difference (to be detected) of 0.5 with expected standard-deviation of difference = 0.5, correlation coefficient of 0.5, a= 5% (two-sided) for a power greater than 90% (1-β=97%).

Subjects are included after a screening visit (visit 0), during which routine laboratory biochemical tests are performed, an electrocardiogram is taken, blood pressure, weight and height are measured; physical examination including testis evaluation and semen parameters are analyzed according to WHO standards 1999 .

The subjects take atorvastatin orally (10mg/day (d), Tahor©, Pfizer Laboratory) during 5 months allowing to study atorvastatin effects on human spermatogenesis and epididymal maturation (one cycle requiring approximately 3 months).

Blood and semen parameters were measured :

* before to take atorvastatin treatment (visit 1)
* at the end of the therapy (visit 3)
* and 3 months after the end of treatment, (visit 4) to perform measurements during different cycles of spermatogenesis on a same subject. After two months of treatment, a consultation (visit 2) is realized to ensure good tolerance to treatment and to control treatment efficiency.

Biochemical clinical and semen measurements take before treatment were considered as "control baseline measures".

ELIGIBILITY:
Inclusion Criteria:

* Men :
* between 18 and 65 years ;
* with normal conventional semen parameters and negative semen culture according to WHO standards 1999 : volume ejaculate ≥ 2 ml, sperm count ≥ 20millions/ml, total motility ≥ 50% progressive motility ≥ 30%, typical forms ≥ 20%;
* with normal blood lipid profile: total cholesterol < 2.50g/L, triglycerides < 1.70g/L, HDL-C > 0.35 g/L and LDL-C < 2.2 g/L;
* without known pathology or ongoing treatment

Exclusion Criteria:

* Subjects with medical or surgical history that may make them at risk during the study,
* Subjects with cons-indications to taking atorvastatin
* Subjects with an active liver disease or increased level of serum transaminases
* Subjects with a history of allergy
* Subjects whose lipid parameters do not match the inclusions criteria or receiving lipid-lowering therapy
* Subject with abnormal semen analysis or cryptorchidism or a varicocele
* Subjects who participated in another clinical trial or other experimentation or other tolerance study of a drug

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Observations of all modifications on semen quality after 5 months of atorvastatin treatment | at month 5
Observations of all modifications on semen quality after 5 months of atorvastatin treatment and after 3 months after its withdrawal | at month 8

SECONDARY OUTCOMES:
hormonal profile: gonadotropins and total testosterone plasma levels | at month 5
  All modifications observed after 5 months of atorvastatin therapy and after 3 months after the end of treatment on
lipid composition of sperm and seminal fluid | at month 5
  All modifications observed after 5 months of atorvastatin therapy and after 3 months after the end of treatment on
spermatozoa capacitation markers | at month 5
  All modifications observed after 5 months of atorvastatin therapy and after 3 months after the end of treatment on
accessory glands markers | at month 5
  All modifications observed after 5 months of atorvastatin therapy and after 3 months after the end of treatment on

CONTACTS AND LOCATIONS:
Overall Officials: Igor TAUVERON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pons-Rejraji H, Brugnon F, Sion B, Maqdasy S, Gouby G, Pereira B, Marceau G, Gremeau AS, Drevet J, Grizard G, Janny L, Tauveron I. Evaluation of atorvastatin efficacy and toxicity on spermatozoa, accessory glands and gonadal hormones of healthy men: a pilot prospective clinical trial. Reprod Biol Endocrinol. 2014 Jul 12;12:65. doi: 10.1186/1477-7827-12-65. PMID 25016482